CLINICAL TRIAL: NCT02838979
Title: Randomized Cross-over Trial of Oral L-Glutamine vs Maltodextrin on Mitochondrial Function in Chronic Kidney Disease
Brief Title: Trial of Oral Glutamine on Mitochondrial Function in CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: New York Medical College (Other); Emory University (Other); Vanderbilt University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jonathan Himmelfarb, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 47861; 5K23DK099442 (NIH)
Record Dates: First submitted 2016-07-08; First posted 2016-07-20 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Disease; Sarcopenia; Endothelial Dysfunction; Muscle Mitochondrial Function; Kidney Disease
Keywords: Glutamine; Chronic Kidney Disease
MeSH Terms: conditions — Cardiovascular Diseases; Sarcopenia; Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral L-Glutamine first, then Maltodextrin (Experimental): Subjects will receive 0.4 g/kg/day of L-glutamine (Nutrestore, EMMAUS Life Sciences, Inc Torrance, CA) in three divided daily doses OR identical appearing maltodextrin powder.
  Duration 2 weeks
  Interventions: Dietary Supplement: First Intervention (14 days); Other: Washout (3 weeks); Dietary Supplement: Second Intervention (14 days)
- Maltodextrin first, then L-glutamine (Experimental): Subjects will crossover to receiving the study product which they did not receive in the first period.
  Either 0.4 g/kg/day of L-glutamine in three divided daily doses OR identical appearing maltodextrin powder.
  Duration 2 weeks
  Interventions: Dietary Supplement: First Intervention (14 days); Other: Washout (3 weeks); Dietary Supplement: Second Intervention (14 days)

INTERVENTIONS:
Dietary Supplement: First Intervention (14 days) — Oral Glutamine or Maltodextrin for 2 weeks
Other: Washout (3 weeks) — No study product is taken prior to beginning crossover
Dietary Supplement: Second Intervention (14 days) — Oral Glutamine or Maltodextrin for 2 weeks

SUMMARY:
The primary goal of proposed investigation is to study the impact of oral glutamine supplementation on muscle mitochondrial and endothelial cell function measured mitochondrial energetics and vascular function using 31P magnetic resonance spectroscopy and optical spectroscopy (MRS/OS) among persons with moderate-severe CKD. The secondary objective is to describe the impact of oral glutamine supplementation on mitochondrial metabolic profile as well as inflammatory and oxidative stress biomarkers among persons with chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease is associated with endothelial cell dysfunction and muscle wasting contributing to the heightened risk of cardiovascular morbidity, mortality and functional limitation. Accumulation of toxins in renal disease may adversely impact endothelial cell nitric oxide bioavailability and endothelial Nitric Oxide Synthase (eNOS) function consequently heightening oxidative stress and suppressing mitochondrial biogenesis. To date no studies have investigated potential therapies for endothelial and muscle dysfunction in renal disease target mitochondrial metabolic and energetic processes.

Animal studies of uremia underscore mitochondrial dysfunction as a potential precursor for endothelial dysfunction. In particular, uremia has been linked to a proteomic signature indicative of metabolic blockage of TCA cycle activity and fatty acid beta-oxidation. Both of these processes are localized to the mitochondria and may suggest that decreased mitochondrial mass or function may augur endothelial dysfunction in renal disease.

Glutamine, an anaplerotic agent and precursor to the antioxidant glutathione, is a potential therapeutic agent bypassing the metabolic block associated with reduced TCA cycle and improving antioxidant reserve. The primary goal of proposed investigation is to study the impact of oral glutamine supplementation on muscle mitochondrial and endothelial cell function measured mitochondrial energetics and vascular function using 31P MRS/OS among persons with moderate-severe CKD. The secondary objective is to describe the impact of oral glutamine supplementation on mitochondrial metabolic profile as well as inflammatory and oxidative stress biomarkers among persons with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 20 and 69 years of age
* Diagnosis of moderate-severe CKD, defined in this study as an estimated glomerular filtration rate (eGFR) of ≤60ml/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration equation
* Ability to understand and provide informed consent to participate in the study

Exclusion Criteria:

* On chronic dialysis
* Expectation to start dialysis within 6 months or dialysis access in place.
* Pregnant
* Have physical immobility (defined by wheelchair use)
* Insulin dependent diabetes
* Have implants incompatible with MRI
* Exercise limiting cardiopulmonary disease (e.g. angina, severe heart valve disease, severe COPD, coronary ischemia)
* Use of anticoagulation (i.e. warfarin)
* Baseline systolic blood pressure >160 or diastolic blood pressure >100
* Inflammatory conditions (e.g. autoimmune disease, HIV)
* Thyroid disease
* Dementia or inability to consent
* Cirrhosis, active/chronic hepatitis
* Use medications interfering with muscle or mitochondrial function, including steroids, anti-psychotic, Coenzyme Q-10, immunosuppresssives, antivirals, and muscle relaxants
* Weight >300 lbs
* Personal history or family history of deep vein thrombosis, pulmonary embolism
* Active malignancy
* Patients hospitalized within the past 60 days for any reason.
* Patients with a history of a major atherosclerotic event (defined as combined incidence of myocardial infarction, urgent target-vessel revascularization, coronary bypass surgery, and stroke) within 3 months

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — Kidney Research Insitute
Locations (1):
- Kidney Research Institute, University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Ziegler TR, Benfell K, Smith RJ, Young LS, Brown E, Ferrari-Baliviera E, Lowe DK, Wilmore DW. Safety and metabolic effects of L-glutamine administration in humans. JPEN J Parenter Enteral Nutr. 1990 Jul-Aug;14(4 Suppl):137S-146S. doi: 10.1177/0148607190014004201. PMID 2119459
- [Background] Amara CE, Marcinek DJ, Shankland EG, Schenkman KA, Arakaki LS, Conley KE. Mitochondrial function in vivo: spectroscopy provides window on cellular energetics. Methods. 2008 Dec;46(4):312-8. doi: 10.1016/j.ymeth.2008.10.001. Epub 2008 Oct 16. PMID 18930151
- [Background] Jones DP, Liang Y. Measuring the poise of thiol/disulfide couples in vivo. Free Radic Biol Med. 2009 Nov 15;47(10):1329-38. doi: 10.1016/j.freeradbiomed.2009.08.021. Epub 2009 Aug 26. PMID 19715755

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral L-Glutamine First, Then Maltodestrin: Subjects will receive 0.4 g/kg/day of L-glutamine (Nutrestore, EMMAUS Life Sciences, Inc Torrance, CA) in three divided daily doses. Duration 2 weeks
  L-glutamine: Oral Glutamine for 2 weeks at dose of 0.4mg/kg/day in three divided daily doses
- Maltodextrin First, Then L-glutamine: Identical appearing maltodextrin powder.
  Maltodextrin: Oral maltodextrin as described for the active agent: 2 weeks at dose of 0.4mg/kg/day in three divided daily doses.
Period: Overall Study
Arm/Group | Oral L-Glutamine First, Then Maltodestrin | Maltodextrin First, Then L-glutamine
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- L-Glutamine First, Then Maltodextrin: Subjects will first receive 0.4 g/kg/day of L-glutamine (Nutrestore, EMMAUS Life Sciences, Inc Torrance, CA) first, then crossover taking Maltodextrin.
- Maltodextrin First, Then L-glutamine: Subjects will first receive Identical appearing maltodextrin powder first, then crossover to taking L-glutamine.
- Total: Total of all reporting groups
Arm/Group | L-Glutamine First, Then Maltodextrin | Maltodextrin First, Then L-glutamine | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (16.6) | 58 (9.8) | 58 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Muscle Mitochondrial Function
Description: 31P MRS/OS was used to measure mitochondrial phosphorylation capacity (ATPmax).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mM ATP/s
Groups:
- L-Glutamine: L-glutamine: Oral Glutamine for 2 weeks at dose of 0.4mg/kg/day in three divided daily doses
- Maltodextrin: Identical appearing maltodextrin powder.
  Maltodextrin: Oral maltodextrin as described for the active agent: 2 weeks at dose of 0.4mg/kg/day in three divided daily doses.
Arm/Group | L-Glutamine | Maltodextrin
Number analyzed (Participants) | 11 | 11
mM ATP/s | 0.88 (0.30) | 0.90 (0.34)
Statistical Analysis 1: Comparison: L-Glutamine vs Maltodextrin; Test type: Superiority; p = 0.15, ANOVA — P-value for the interaction of treatment and sequence; Two-way ANOVA was used to assess differences between the groups; Mean Difference (Final Values) = -0.01, Standard Deviation 0.34

2. Secondary Outcome: Change in Force-time Integral Area Under the Curve in Active Agent vs. Placebo
Description: To test if glutamine improves objective isometric muscle fatigue by comparing the measurement of FTI from each arm. Muscle fatigability was tested by calculating FTI as the area under the force-time curve during isometric force generated at 70 % of maximal voluntary contraction (MVC),
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: N*s
Arm/Group | L-Glutamine | Maltodextrin
Number analyzed (Participants) | 11 | 11
N*s | 58.87 (24.07) | 52.36 (21.22)
Statistical Analysis 1: Comparison: L-Glutamine vs Maltodextrin; Test type: Superiority; p = 0.86, ANOVA — P-value for the interaction of treatment and sequence; Two-way ANOVA was used to assess differences between the groups; Mean Difference (Final Values) = -7.39, Standard Deviation 22.18

3. Secondary Outcome: Muscle Fatigue
Description: To test the effect of glutamine supplementation on muscle endurance, sum of the muscle force (force-time integral, FTI, N*s) normalized to maximum voluntary contraction (MVC, N) generated during voluntary contraction.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: s-1
Arm/Group | L-Glutamine | Maltodextrin
Number analyzed (Participants) | 11 | 11
s-1 | 2.52 (1.09) | 2.41 (1.03)
Statistical Analysis 1: Comparison: L-Glutamine vs Maltodextrin; Test type: Superiority; p = 0.44, ANOVA — P-value for the interaction of treatment and sequence; Two-way ANOVA was used to assess differences between the groups; Median Difference (Final Values) = -0.10, Standard Deviation 1.04

4. Other Pre Specified Outcome: Plasma NAD+ Levels
Description: To test if glutamine improves plasma NAD+ compared to placebo. Plasma NAD+ concentrations were quantified in mM using 31p MRS based in vivo assay.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | L-Glutamine | Maltodextrin
Number analyzed (Participants) | 11 | 11
mM | 0.95 (0.25) | 0.98 (0.19)
Statistical Analysis 1: Comparison: L-Glutamine vs Maltodextrin; Test type: Superiority; p = 0.36, ANOVA — P-value for the interaction of treatment and sequence; Two-way ANOVA was used to assess differences between the groups; Mean Difference (Final Values) = 0.06, Standard Deviation 0.21

5. Post Hoc Outcome: Maximal Voluntary Contraction
Description: To test if glutamine improves maximal voluntary contraction compared to placebo. Maximum voluntary contraction (MVC) was determined by the isometric force generated using first dorsal interosseous (FDI) muscle against a force transducer.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: N/m
Arm/Group | L-Glutamine | Maltodextrin
Number analyzed (Participants) | 11 | 11
N/m | 23.6 (6.834) | 23.22 (8.967)
Statistical Analysis 1: Comparison: L-Glutamine vs Maltodextrin; Test type: Superiority; p = 0.60, ANOVA — P-value for the interaction of treatment and sequence; Two-way ANOVA was used to assess differences between the groups; Mean Difference (Final Values) = -0.45, Standard Deviation 7.87

ADVERSE EVENTS:
Time Frame: 7 weeks
Groups:
- Maltodextrin: Identical appearing maltodextrin powder.
Arm/Group | L-Glutamine | Maltodextrin
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT02838979/Prot_SAP_000.pdf
  • Informed Consent Form (2016-03-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT02838979/ICF_001.pdf